CLINICAL TRIAL: NCT00384488
Title: Effectiveness of Automated Telephone Intervention on Behavioral and Weight Outcomes for Patients With Pre-Diabetes.
Brief Title: Automated Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CO-04PEsta-02
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Pre-Diabetes
Keywords: Diabetes mellitus; Weight control; Healthy eating; Physical Activity
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Motor Activity

INTERVENTIONS:
Behavioral: Interactive Voice Response System (IVR)

SUMMARY:
The objective for this pilot project is to determine the feasibility and effectiveness of the Interactive Voice Response protocol (IVR) on physical activity and eating behaviors in a group men and women who have been identified by their physician as being pre-diabetic. We hypothesize that participants receiving the IVR follow-up will have greater positive changes in their physical activity and eating behaviors when compared to those who receive only the standard-care pre-diabetes class.

DETAILED DESCRIPTION:
Patients diagnosed with pre-diabetes present a unique opportunity for health care providers to implement preventive practices. Behavioral intervention strategies that target weight reduction or maintenance and increased fitness not only provide exceptional cardiovascular benefits, but also play an important role in delayed development or prevention of type 2 diabetes mellitus (DM). This study was designed to determine the feasibility and effectiveness of automated telephone support calls targeting physical activity and healthful eating as strategies for weight loss for patients with pre-diabetes.

Participants with pre-diabetes who participated in a 90-minute diabetes prevention class were consented to participate in this behavioral study and were then randomly assigned to receive automated telephone support targeting physical activity and nutrition weight loss strategies or to a no-contact control group. Objective physical activity (accelerometer), self-reported dietary intake, and body weight were assessed at baseline and at 3-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Kaiser-Permanente of Colorado members age 18 and above who have been diagnosed with pre-diabetes and who have enrolled in a clinically indicated pre-diabetes class.
* Subjects must be English speaking and have a telephone

Exclusion Criteria:

Pregnant females

* Enrollment in another research study involving diabetes or weight management during the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2004-05; Study Completion 2006-05

PRIMARY OUTCOMES:
Weight loss

SECONDARY OUTCOMES:
Increased physical activity
Improved healthy eating habits
Weight maintenance
Reduction in progression to type 2 DM

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Estabrooks, PhD, Principal Investigator — Kaiser-Permanente of Colorado Clinical Research Unit
Locations (1):
- Kaiser-Permanente of Colorado, Aurora, Colorado, United States